CLINICAL TRIAL: NCT02823288
Title: Refinement and Evaluation of a Multilevel Intervention for Preventing Men's Use of Violence in Urban South Africa (Sonke CHANGE Trial)
Brief Title: Multilevel Intervention for Preventing Men's Use of Violence in Urban South Africa (Sonke CHANGE Trial)
Acronym: Sonke CHANGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: Sonke Gender Justice (Unknown); Medical Research Council, South Africa (Other); Department for International Development, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Abigail Hatcher, Senior Researcher, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: M150443
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Domestic Violence; Sexual Assault and Rape; Masculinity
Keywords: intimate partner violence; masculinity; community mobilization; social intervention; rape
MeSH Terms: conditions — Masculinity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sonke CHANGE intervention condition (Experimental): This arm (n=9 clusters) will receive the Sonke CHANGE intervention for 12 months.
  Interventions: Other: Sonke CHANGE intervention
- Control condition (No Intervention): In this arm (n=9 clusters), no activities will take place during the trial period outside of data collection.

INTERVENTIONS:
Other: Sonke CHANGE intervention — The Sonke CHANGE intervention is a multi-level model aimed at individual, group, community, and societal levels. Sonke's programming is comprised of three core components:
  1. Workshops based on the premise that deeply held gender and sexuality beliefs can be critically examined and transformed in a reflective group setting. Workshops aim to challenge inequitable and harmful ideas about manhood and encourage men to take action to promote equality.
  2. Community Action Teams (CATs) are comprised of interested men and women, who mobilize on a voluntary basis around issues in their neighborhoods. Methods include ambush theatre, murals painting, door to door campaigns, street soccer festivals, rallies, and community dialogues.
  3. Local Advocacy is undertaken by CAT members, who aim to hold government and other duty bearers to account for VAWG prevention. CAT members join local community structures to advance community education and local government accountability.
  Arms: Sonke CHANGE intervention condition

SUMMARY:
South Africa has one of the highest rates of violence towards women globally. However, little is known about how to prevent men's use of violence. The Sonke CHANGE Trial tests an intervention that targets men as individuals, groups, and community members in a peri-urban setting in South Africa. Eighteen neighborhoods will be randomly assigned to either the intervention condition or a control group. By speaking to men at baseline, 12 months, and 24 months, investigators will learn whether violence and other health behaviors shift over time. Alongside the trial, qualitative research will explore how the intervention took place and why participants may change attitudes or behaviors.

DETAILED DESCRIPTION:
This study will refine and evaluate a multi-level model for reducing violence against women and girls in urban South Africa.

The intervention is a refinement of an existing gender-transformative programme that includes community mobilisation and advocacy. Called the Sonke CHANGE intervention, it will extend beyond a conventional group-based workshop approach to address the multi-level nature of violence and create an enabling environment for men to embrace more equitable forms of masculinity. Given the strong associations between masculinities and men's use of partner violence, now is an opportune moment to test the Sonke CHANGE model to determine its impact on men's use of violence.

The multi-level Sonke intervention will be evaluated using a cluster randomised controlled trial design. In a peri-urban setting of Diepsloot, neighbourhood "clusters" (n=18) will be randomly assigned to receive the intervention or a wait-list condition. Baseline, 12 month, and 24 month measures will assess changes in primary outcomes (men's reported use of intimate partner and non-partner violence) and secondary outcomes (severe violence, masculinity norms, harmful alcohol use, mental health). Formative qualitative research will explore the environmental context of Diepsloot, community views on violence, men's mobility, and their experiences of fathering. A longitudinal process evaluation will explore intervention delivery, unfolding of the advocacy element of Sonke CHANGE intervention, and potential mechanisms to change amongst participants.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 40 years of age (inclusive)
* lives in a trial cluster
* willing to participate on basis of written, informed consent

Exclusion Criteria:

* younger than 18 years or older than 40 years
* lives outside of a trial cluster
* unwilling to participate or sign written, informed consent

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2603 (Actual)
Dates: Start 2016-02; Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change in intimate partner violence | 12 months, 24 months
  Men's use of violence towards an intimate partner will be measured using an adapted version of the questionnaire from the South African Medical Research Council's Study on Men's Health and Relationships (6, 61). The questionnaire includes items around emotional abuse, economic abuse, physical violence, and sexual violence. Primary outcomes will be defined as dichotomous outcomes: any use of physical violence and / or any use of sexual violence.

SECONDARY OUTCOMES:
Change in severe violence | 12 months, 24 months
  Men's use of severe violence is defined as any instance of men reporting more than once response to a single physical or sexual IPV item OR a response of once or more than once to two or more physical and/or sexual items.
Change in controlling behavior | 12 months, 24 months
  Male Controlling Behaviour will be measured using the Pulerwitz Sexual Relationship Power and Control scale items (65). This scale has been validated in South Africa (66), and has been used by members of our team in previous studies (67).
Change in gender attitudes | 12 months, 24 months
  Gender Attitudes will be measured using the Gender Equitable Men's Scale (GEM Scale) (63), an 18-item Likert scale. Gender Norms will be comprised of similar items, but phrased in a Likert scale for whether a man's friends hold those beliefs.
Change in harmful alcohol use | 12 months, 24 months
  Harmful alcohol use will be measured using the Alcohol Use Disorders Identification Test (AUDIT), a 10-item scale designed to measure alcohol consumption and identify risks for alcohol abuse and dependence (62).

CONTACTS AND LOCATIONS:
Overall Officials: Nicola J Christofides, PhD, Principal Investigator — University the Witwatersrand
Locations (1):
- Wits School of Public Health, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be available 5 years after the end of the research through an institutional repository managed by the South African MRC. Data sharing will be managed through an application process, whereby the original investigators will be invited to participate in future papers.

REFERENCES:
- [Derived] Hatcher AM, Neilands TB, Rebombo D, Weiser SD, Christofides NJ. Food insecurity and men's perpetration of partner violence in a longitudinal cohort in South Africa. BMJ Nutr Prev Health. 2022 Feb 7;5(1):36-43. doi: 10.1136/bmjnph-2021-000288. eCollection 2022. PMID 35814730
- [Derived] Gibbs A, Dunkle K, Mhlongo S, Chirwa E, Hatcher A, Christofides NJ, Jewkes R. Which men change in intimate partner violence prevention interventions? A trajectory analysis in Rwanda and South Africa. BMJ Glob Health. 2020 May;5(5):e002199. doi: 10.1136/bmjgh-2019-002199. PMID 32424011
- [Derived] Christofides NJ, Hatcher AM, Rebombo D, McBride RS, Munshi S, Pino A, Abdelatif N, Peacock D, Levin J, Jewkes RK. Effectiveness of a multi-level intervention to reduce men's perpetration of intimate partner violence: a cluster randomised controlled trial. Trials. 2020 Apr 25;21(1):359. doi: 10.1186/s13063-020-4185-7. PMID 32334615
- [Derived] Christofides NJ, Hatcher AM, Pino A, Rebombo D, McBride RS, Anderson A, Peacock D. A cluster randomised controlled trial to determine the effect of community mobilisation and advocacy on men's use of violence in periurban South Africa: study protocol. BMJ Open. 2018 Mar 23;8(3):e017579. doi: 10.1136/bmjopen-2017-017579. PMID 29574438
- See also: Study Design Brief — http://www.genderjustice.org.za/publication/one-man-can-randomised-control-trial-in-diepsloot-johannesburg/
- See also: Evidence Brief: Baseline Findings — http://www.whatworks.co.za/resources/project-resources/item/301-sonke-change-trial-evidence-brief